CLINICAL TRIAL: NCT05961436
Title: Pericapsular Nerve Group (PENG) Block Versus Femoral Nerve Block: Impact on Quadriceps Muscle Strength in Patients With Hip Fracture - a Prospective Randomized Controlled Trial
Brief Title: Comparing PENG and Femoral Nerve Blocks in Patients With Hip Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Dina Mahmoud Fakhry, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Management, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMBSUREC/06062023/Fakhry
Record Dates: First submitted 2023-07-11; First posted 2023-07-27 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Pain
Keywords: Femoral nerve; Pericapsular nerve group; Pain; Hip fracture
MeSH Terms: conditions — Pain; Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG block group (Active Comparator): using ultrasound-guided technique, a total of 20ml of 0.25 % bupivacaine will be injected after negative aspiration.
  Interventions: Procedure: PENG block
- FN block group (Active Comparator): using ultrasound-guided technique, after negative aspiration, 20 mL of 0.25 % bupivacaine will be administered.
  Interventions: Procedure: FN block

INTERVENTIONS:
Procedure: PENG block — Using ultrasound-guided technique, a total of 20ml of 0.25 % bupivacaine will be injected after negative aspiration.
  Arms: PENG block group
Procedure: FN block — Using ultrasound-guided technique, after negative aspiration, 20 mL of 0.25 % bupivacaine will be administered.
  Arms: FN block group

SUMMARY:
The aim of this work is to compare between the use of PENG block and femoral nerve block for perioperative pain management in patients with hip fracture.

DETAILED DESCRIPTION:
Hip fractures are common orthopaedic problem especially in elderly population which is associated with significant morbidity and mortality. Early surgical reduction and fixation is the preferred treatment in most patients. Significant pain, if inadequately controlled, can impair early rehabilitation and functional recovery and can reduce patient satisfaction after surgery . Combinations of systemic analgesics, intra-articular injection, and neuraxial and peripheral nerve blocks should be considered as the integral components of the perioperative pain management plan. Among these, intra-articular local anaesthetic injections have been shown to play a potential role in providing analgesia after hip arthroplasty. The risks of this procedure include hematoma, nerve damage, local anaesthetics toxicity, intravenous injection of local anesthetics and septic osteoarthritis, but their occurrence is very rare. Several peripheral nerve blocks, including fascia iliaca block, femoral block (FB), and some interfascial plane blocks such as quadratus lumborum block (QLB), have also been suggested to decrease postoperative pain and opioid use. Lumbar plexus block/psoas compartment block is a technically difficult deep block that requires greater skill and hence can be time consuming. The lumbar paravertebral region is highly vascular and non-compressible. Hence, patients on anti-coagulation are at high risk for bleeding complications. There is also high risk of unintentional neuraxial block or inadvertent intravascular injection with local anaesthetic systemic toxicity. Some nerve branches responsible for hip joint innervation may not be blocked by QLB, which should be taken into consideration while using these blocks for hip fracture. High-volume suprainguinal fascia iliaca block and traditional fascia iliaca block have also been reported to be associated with a significant incidence of muscle weakness and to predispose the patient to fall. The anterior hip capsule is innervated by the obturator nerve (ON), accessory obturator nerve (AON), and femoral nerve (FN) as reported by previous anatomic studies. The anterior capsule is the most richly innervated section of the joint, suggesting these nerves should be the main targets for hip analgesia. Femoral block (FB) does not block the AON or the articular branches of the ON. Also, femoral nerve block accompanied by decreasing the strength of quadriceps muscles. Pericapsular nerve group (PENG) block was described in 2018 and reported that it was successfully used for postoperative pain management in hip surgery. The PENG block is a technique that involves deposition of local anaesthetic in the musculofascial plane between the psoas muscle and the superior pubic ramus for the blockade of the articular branches of the FN, ON and AON that provide sensory innervation to the anterior hip capsule.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a hip fracture.
* Aged 50 years and older.

Exclusion Criteria:

* Consent refusal.
* Allergy to local anaesthetics.
* Infection of the puncture site.
* Dementia or cognitive impairment.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Quadriceps muscle strength in recovery. | 24 hours of the procedure
  Quadriceps muscle strength will be assessed using Oxford muscle strength grading with grouped scores of intact (5/5), reduced (1-4/5) and absent (0/5).
  Muscle Grading Scores:
  0 No detectable muscle contraction (visible or palpation)
  1. Detectable contraction (visible or palpation), but no movement achieved
  2. Limb movement achieved, but unable to move against gravity
  3. Limb movement against resistance of gravity
  4. Limb movement against gravity and external resistance
  5. Normal strength

SECONDARY OUTCOMES:
Visual analogue scale | 24 hours of the procedure.
  before and 30 minutes after the block both at rest and during dynamic hip movement.
  0 means no pain 10 means the worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Dina M Fakhry, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-Suef University hospital, Banī Suwayf, Beni Suweif Governorate, Egypt